CLINICAL TRIAL: NCT00200642
Title: Evaluation of the Efficiency of Radiofrequency in the Treatment of Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/03/6-F
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux. PPI. Radiofrequency
MeSH Terms: conditions — Gastroesophageal Reflux

INTERVENTIONS:
Device: Stretta® System

SUMMARY:
Gastroesophageal reflux disease is a frequent disease and which heavily affects the patients' quality of life. To alleviate symptoms and ease the healing of lesion, patients very often need to continuously take anti-secretory drugs (Proton pump inhibitors or PPIs), which, despite their efficiency, do not cure the disease. For these PPI dependent patients, an anti-reflux surgery (fundoplication often made by coelioscopy) is a possible alternative but it has a significant morbidity rate and even an estimated post-operative mortality of 0.8% outside of expertise centres. Therefore, new therapeutic endoscopic approaches, supposed to be less invasive and less expensive than surgery have been developed during the last three years. Among them, radiofrequency (Stretta® procedure) consists in administering a high frequency current in the cardia area, in order to induce thanks to a thermal effect a sub-mucous remodelling and a modification of the compliance of the cardia regionThe aim of this project carried out in 8 French centres and 2 European centers is to assess through a randomised trial, the efficiency of radiofrequency on PPI dependent patients. The study will be carried out in 2 phases with patients who have been fully informed of the project statement, and particularly of the potential risks of the radiofrequency technique and have given their written acceptation to participate to the study.The first phase, which will last 6 to 11 weeks, will aim at making sure that patients are PPI dependent and define their needs. After this initial phase, patients will be randomised between those who will carry on with the PPI treatment or the radiofrequency treatment. The follow up after this randomisation will last one year. The first assessment of the therapeutic efficiency will be done at 6th month. The 6 additional follow up months will be required for the assessment of mid-term side effects of the treatment and the rate of symptomatic recurrences.

ELIGIBILITY:
Inclusion Criteria:

1. Patient above 18 years old
2. Suffering from typical symptoms of reflux (heartburn and/or acid regurgitation and/or epigastric burns with ascending radiations)
3. Symptoms occurring at least 3 times a week without treatment
4. Symptoms disappearing under full doses PPI treatment
5. Requiring a continuous treatment for more than 3 months to get rid of symptoms (or nearly)
6. Total consent signed from patient

Exclusion Criteria:

1. Contraindications to the radiofrequency technique:

   * Columnar lined oesophagus ³ 3 cm height
   * Barret's mucosa presenting dysplasia
   * History of treated columnar lined oesophagus
   * Hiatus hernia with a size over 3 cm
   * History of Stage C or D esophagitis in the Los Angeles classification (18), or in progress
   * History of oesophageal stenosis
   * History of gastric or oesophageal surgery
   * Presence of oesophageal and/or cardial varicose veins
   * Presence of a cardiac pacemaker or implanted defibrillator (when confirmed by the manufacturer that use of RF energy will not interfere, it's ok to do patients!)
   * Impossibility to interrupt a anticoagulant treatment or serious disorders of haemostasis
2. General contraindications:

   * Contraindication to general anaesthesia
   * Existence of an associated serious disease making fear that the patient will live less than a year
   * Incapacity to understand and sign a sensible consent of participation to the study
   * Chronic alcoholism defined by a daily consumption of alcohol over 60 g
   * Morbid obesity defined by a rate of body mass higher that 35
   * Patients suffering from atypical GERD symptoms (especially extra-digestive) will not be included in the study if these symptoms are not associated with typical reflux symptoms (heartburn or regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The main endpoint will be the possibility or not to stop the PPI treatment (or to reduce the dose by at least 50%), 6 months after administering (or not) just one radiofrequency session.

SECONDARY OUTCOMES:
The evaluation of tolerance,
the description of potential complications entailed by the technique and the measure of GERD recurrence rate on patients over a one-year period.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Galmiche, MD, Principal Investigator — Nantes UH
Locations (1):
- Nantes University Hospital, Nantes, France